CLINICAL TRIAL: NCT05331014
Title: A Multi-center, Randomized, Double-blind, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0101+C2101 in Patients With Dyslipidemia and Hypertension.
Brief Title: To Evaluate the Efficacy and Safety in Patients With Dyslipidemia and Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JWP-PVA-301
Record Dates: First submitted 2022-04-04; First posted 2022-04-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dyslipidemia; Hypertension
MeSH Terms: conditions — Dyslipidemias; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JW0101+C2101 (Experimental): LivaloVA
  Interventions: Drug: LivaloVA
- JW0101+C2102 (Active Comparator): LivaloV
  Interventions: Drug: LivaloV
- C2101 (Active Comparator): VA
  Interventions: Drug: VA

INTERVENTIONS:
Drug: LivaloVA — For 8 weeks(PO, QD)
  Other Names: JW0101+C2101
  Arms: JW0101+C2101
Drug: LivaloV — For 8 weeks(PO, QD)
  Other Names: JW0101+C2102
  Arms: JW0101+C2102
Drug: VA — For 8 weeks(PO, QD)
  Other Names: C2101
  Arms: C2101

SUMMARY:
A Multi-center, Randomized, Double-blind, Parallel, phase III Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0101+C2101 in Patients with Dyslipidemia and Hypertension.

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, parallel-design, phase III clinical study

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and dyslipidemia

Exclusion Criteria:

* The subject not meet the specified msBP and LDL-C level

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
msSBP (8 weeks) lowering effect, LDL-C (8 weeks) lowering effect | week 8
  change in msSBP and LDL-C level

SECONDARY OUTCOMES:
efficacy and safety | week 8
  change in msSBP and LDL-C level

CONTACTS AND LOCATIONS:
Overall Officials: Gyurok Han, CI, Principal Investigator — Gangdong Sacred Heart Hospital
Locations (1):
- Gangdong Sacred Heart Hospital, Seoul, Korea, South Korea